CLINICAL TRIAL: NCT03307278
Title: Effects and Mechanism of House Dust Mite Induced Inflammasome Activation on Corticosteroid Resistance
Brief Title: House Dust Mite Induced Inflammasome Activation on Corticosteroid Resistance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The research project cannot be implemented because the project has not received funding subsidies
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH106-REC3-115
Record Dates: First submitted 2017-09-26; First posted 2017-10-11 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — Antigens, Dermatophagoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Steroid resistance in HDM allergic patients (Experimental)
  Interventions: Biological: House dust mite
- Steroid resistance in non HDM allergic subjects (Experimental)
  Interventions: Biological: House dust mite

INTERVENTIONS:
Biological: House dust mite — As a stimulant to induce inflammasome activation

SUMMARY:
In this project, PBMCs will be isolated from HDM allergic and non allergic patient and then stimulated with HDM crude extract. The expression of inflammasome and the correlation of inflammasome activation and steroid resistance will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* HDM allergic and non allergic subjects

Exclusion Criteria:

* Pregnant subject, cancer

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-11-30 (Estimated); Primary Completion 2018-09-06 (Estimated); Study Completion 2018-09-06 (Estimated)

PRIMARY OUTCOMES:
inflammasome activation by HDM | 6 hours
  The expression of NLRP3 in PBMCs will be measured by western blot after HDM stimulation.
Steroid receptor phosphorylation by HDM | 6 hours
  The expression of steroid receptor will be detected by western blot and real-time PCR after HDM stimulation.

IPD SHARING:
Plan to Share IPD: Undecided